CLINICAL TRIAL: NCT00161954
Title: Open Phase IV Clinical Study to Evaluate the Immunogenicity and Safety of a Rapid Immunization Schedule With FSME-IMMUN 0.5 mL in Healthy Adults Aged 16 - 65 Years
Brief Title: Immunogenicity and Safety Study of a Rapid Immunization Schedule With FSME-IMMUN 0.5 mL in Healthy Adults Aged 16 - 65 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 225
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
Keywords: Tick-Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The objective of this study is to establish the earliest time point at which vaccines are expected to show seropositive antibody levels after vaccination with FSME-IMMUN 0.5 mL using a rapid immunization schedule (2 vaccinations administered 12 +/- 2 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Understanding the nature of the study, agreement to its provisions and written informed consent
* Written informed consent of subject´s parents / legal guardians (if subject is under 18 years of age)
* Aged >= 16 years (from the 16th birthday) to <= 65 years (to the last day before the 66th birthday)
* Clinically healthy, (i. e. the physician would have no reservations vaccinating with FSME-IMMUN 0.5 ml outside the scope of a clinical trial)
* Negative pregnancy test result at the first medical examination (if female and capable of bearing children)
* Agreeing to employ adequate birth control measures for the duration of the study (if female and capable of bearing children)
* Agreeing to keep a subject diary.

Exclusion Criteria:

* History of any previous TBE vaccination
* History of TBE infection
* History of infection with other flaviviruses
* History of vaccination against yellow fever and/or Japanese B-encephalitis
* History of allergic reactions, in particular to one of the components of the vaccine
* Suffering from a disease (e.g. autoimmune disease) or undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions
* Known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages)
* Donation of blood or plasma within one month of study start
* Having received a blood transfusion or immunoglobulins within one month of study entry
* HIV positivity (an HIV test is not required specifically for the purpose of this study
* Simultaneous participation in another clinical trial including administration of an investigational product
* Participating in any other clinical study within six weeks prior to study start
* Participated in another Baxter vaccine study within the last six months (with the exception of follow-up studies)
* Pregnancy or lactation (if female)
* Having received any other vaccination within two weeks prior to study entry

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-03; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter BioScience
Locations (1):
- SGS Biopharma Research Unit Stuivenberg, Antwerp, Belgium

REFERENCES:
- [Derived] Orlinger KK, Hofmeister Y, Fritz R, Holzer GW, Falkner FG, Unger B, Loew-Baselli A, Poellabauer EM, Ehrlich HJ, Barrett PN, Kreil TR. A tick-borne encephalitis virus vaccine based on the European prototype strain induces broadly reactive cross-neutralizing antibodies in humans. J Infect Dis. 2011 Jun 1;203(11):1556-64. doi: 10.1093/infdis/jir122. PMID 21592984